CLINICAL TRIAL: NCT01536119
Title: Evaluating the Effectiveness of a Coparenting Breastfeeding Support Intervention on Exclusive Breastfeeding Rates at 12 Weeks Postpartum
Brief Title: Evaluating a Coparenting Breastfeeding Support Intervention
Acronym: COSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Cindy-Lee Dennis, Associate Professor, Lawrence S. Bloomberg Faculty of Nursing, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27286
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Parenting; Breastfeeding
Keywords: Breastfeeding; Coparenting; Infant feeding; Fathers' support; Breastfeeding support; Breastfeeding support intervention; clinical trial
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coparenting Breastfeeding Support Intervention (Experimental): The intervention group will receive a in-hospital discussion, a video, a workbook,a breastfeeding booklet, access to a secure study website, two follow-up emails, and one telephone call.
  Interventions: Behavioral: Coparenting Breastfeeding Support Intervention
- Usual Care Group (No Intervention): The usual care group will receive standard postpartum care in the hospital and in the community

INTERVENTIONS:
Behavioral: Coparenting Breastfeeding Support Intervention — The intervention group will receive standard care offered to breastfeeding women in the hospital and community with the addition of a multifaceted coparenting breastfeeding support intervention, which will include an in hospital discussion, a video, workbook, breastfeeding booklet, and access to a secure website. Additionally, two follow-up phone calls will be made at 1 and 4 weeks postpartum. This intervention has been designed with coparenting elements and contains extensive breastfeeding information.
  Other Names: Other Names:; Coparenting Group
  Arms: Coparenting Breastfeeding Support Intervention

SUMMARY:
The purpose of this trial is to evaluate the effectiveness of a Coparenting Breastfeeding Support Intervention with first time parents on exclusive breastfeeding rates at 12 weeks postpartum. Partner support and the coparenting relationship will also be evaluated.

DETAILED DESCRIPTION:
Breastfeeding is the recommended infant feeding method by leading health authorities. This recommendation is based on the many health benefits breastfeeding provides to both women and their infants. Breastfeeding rates in Canada, however, are suboptimal, with nearly half of mothers discontinuing exclusive breastfeeding in the first three months and less than twenty-five percent of mothers meeting the recommendation of exclusive breastfeeding to six months.

There are many factors associated with the premature cessation of exclusive breastfeeding. They include demographic, biological, psychosocial, and social factors. Some of these factors are not modifiable, such as age, social status, and education level, as they are not amenable to an intervention. One possible modifiable factor, which may assist women in overcoming breastfeeding difficulties, is fathers' support with breastfeeding. Fathers' favourable attitude and support of breastfeeding positively impacts breastfeeding initiation, duration, and exclusivity. Research on ways to assist fathers in providing support for breastfeeding is needed. The ways in which fathers can provide effective support can best be determined through intervention studies designed to increase fathers' supportive behaviour towards breastfeeding. Specifically, a coparenting framework to guide such interventions would be optimal as coparenting teaches parents to work in partnership towards positive child health outcomes. The purpose of this proposed randomized controlled trial is to evaluate the effects of a coparenting breastfeeding support intervention, delivered to primiparous breastfeeding mothers and the infants' fathers (the breastfeeding woman's male partner, who is jointly responsible for the child). It is hypothesized that this intervention will increase exclusive breastfeeding at 12 weeks postpartum. The secondary outcomes will be breastfeeding duration, perceived breastfeeding support, and coparenting at 6 and 12 weeks. Paternal breastfeeding self-efficacy and infant feeding attitude will be assessed at 6 weeks postpartum.

Participants will include first-time breastfeeding women and the infants' fathers who have singleton births and full term healthy infants. Eligible parents who consent to participate will be randomized into either the intervention group or the control group. The control group will receive standard postpartum care, which is routine care in the hospital and community related to breastfeeding. The intervention group will receive standard postpartum care, plus a multifaceted support intervention that includes: (1) a professional-based in-hospital visit in the first two days postpartum that uses a take-home workbook, breastfeeding booklet, and video, (2) two follow-up emails in the first and third week postpartum, (3) one telephone call to the mother at two weeks, and (4) access to a secure study website for a three month period. All of the components in this intervention will contain extensive information on coparenting and breastfeeding. Follow-up data will be collected by the method chosen by participants, either by web-based survey or telephone interview. This data will be collected by a research assistant blinded to group allocation and data collection points will be at 6 and 12 week postpartum.

The results of this study will be of interest to health care professionals who work with breastfeeding women and their families, as well as policy makers designing programs to meet the needs of childbearing families.

ELIGIBILITY:
Inclusion Criteria:

* The target population for the study will be all primiparous breastfeeding women on the postpartum unit who meet the following inclusion criteria:

  1. singleton birth (vaginal and cesarean births)
  2. term infant (37-42 weeks gestation)
  3. speaks and reads English
  4. 18 years of age or older
  5. parents living in the same home, father (the breastfeeding woman's male partner) jointly responsible for the infant.

Exclusion Criteria:

* The exclusion criteria will include:

  1. sharing a hospital room with a study participant
  2. infants or maternal medical problems that interfere with breastfeeding (eg. infant with cleft palate or maternal previous breast surgery)
  3. midwifery patient
  4. infant not discharged home with mother
  5. mother is pumping milk but not breastfeeding
  6. mother does not have access to the internet
  7. mother does not have a telephone.
  8. father not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy-Lee Dennis, PhD, Principal Investigator — University of Toronto
Locations (1):
- North York General Hospital, North York, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at on the postpartum unit of a large Toronto hospital between March 26th and July 15th 2012
Pre-assignment Details: Eligibility determined before recruitment into trial.
Period: Overall Study
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Started | 214 ((107*2= 214) (107 mothers and 107 fathers)) | 214 ((107*2=214) (107 mothers and 107 fathers))
Completed | 197 (104 Mothers + 93 fathers = 197 participants 3 mothers + 14 fathers = 17 did not complete the study) | 200 (105 mothers + 95 fathers = 200 participants 2 mothers + 12 fathers = 14 did not complete the study)
Not Completed | 17 | 14
Not completed — Lost to Follow-up | 17 | 14

BASELINE CHARACTERISTICS:
Population: The baseline participants consisted of 214 participants 107*2=214 107 couples per group (107 mothers and 107 fathers).
Groups:
- Total: Total of all reporting groups
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group | Total
Number analyzed (Participants) | 214 | 214 | 428
Age, Categorical [Number; unit: participants] — This is a measure of maternal age only
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 107 | 107 | 214
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of fathers in the study
  years | 33 (5.2) | 33 (5.5) | 33 (5.4)
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of mothers in the study
  years | 30.4 (3.7) | 30.7 (3.8) | 30.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 107 | 107 | 214
Region of Enrollment [Number; unit: participants] — All couples were enrolled in Canada. 214 couples with 107 couples per group
  participants
    Canada | 107 | 107 | 214

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Breastfeeding Rate at 12 Weeks Postpartum
Description: Exclusive breastfeeding will be determined by asking the mother what she has fed her baby in the last 24 hrs and what she usually feeds her baby. This is consistent with the World Health Organizations definition of exclusive breastfeeding and full breastfeeding described by Labbok and Krasovec (1990). This is defined as no food or liquid other than breast milk given to the infant; however, undiluted drops or syrups consisting of vitamins, minerals supplements or medicines are included (Breastfeeding Committee for Canada, 2006; WHO, 2010).
Time Frame: 12 weeks postpartum
Population: Analysis population included only mothers
Measure: Number; unit: percentage of participants
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 104 | 105
percentage of participants | 70 | 63
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Power analysis was conducted to a 15 % increase in exclusive breastfeeding rates (from 52% to 67%) with 80% power and an alpha of 0.05. A 25% attrition rate waas added. 107 couples were needed per group. Intention to treat analysis conducted. Exclusive breastfeeding at 12 weeks; Test type: Superiority or Other; p = 0.27, Chi-squared; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.91 to 1.38]

2. Secondary Outcome: Exclusive Breastfeeding
Description: as for outcome 1
Time Frame: 6 weeks
Population: Analysis population included only mothers
Measure: Number; unit: percentage of participants
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 104 | 102
percentage of participants | 75 | 62
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.09, Chi-squared; Risk Ratio (RR) = 1.19, 95% CI [0.98 to 1.44]

3. Secondary Outcome: Any Breastfeeding
Description: Any breastfeeding was measured by asking the mother what she had fed her infant in the last 24 hours and what she usually feeds her baby. Any breastfeeding indicated the mother was breastfeeding or providing her infant with expressed breastmilk and this included combined feeding with formula. If the mother responded she was only formula feeding this indicated the infant she was not doing any breastfeeding or being fed any breast milk.
Time Frame: 6 weeks
Population: Analysis population included only mothers
Measure: Number; unit: participants
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 104 | 102
participants | 102 | 94
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.06, Fisher Exact; Risk Ratio (RR) = 1.06, 95% CI [1.00 to 1.13]

4. Secondary Outcome: Any Breastfeeding
Description: as for outcome 3
Time Frame: 12 weeks
Population: Analysis population included only mothers
Measure: Number; unit: participants
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 104 | 105
participants | 100 | 92
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 1.10, 95% CI [1.01 to 1.19]

5. Secondary Outcome: Coparenting Relationship
Description: Coparenting is the degree to which parents work together to achieve parenting goals. This will be measured using Feinberg, Brown and Kan (2010) Coparenting Relationship Scale (CRS) Brief Form. There are 14 items in total in this tool. There is a 7 point response scale ranging from 0 - 6. The total score ranges from 0 - 84. Negative items are reversed and the higher scores indicate positive coparenting.
Time Frame: 6 weeks
Population: Analysis population included only mothers who completed the questionnaire at 6 weeks postpartum.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 98 | 91
units on a scale | 73.01 (9.8) | 71.3 (10.6)
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Brief scale used; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Coparenting Relationship
Description: Coparenting is the degree to which parents work together to achieve parenting goals. This will be measured using Feinberg, Brown and Kan (2010) Coparenting Relationship Scale (CRS). There are 35 items in total in this tool. There is a 7 point response scale ranging from 0 to 6. Total scores range from 0 - 210. Negative items are reversed. Higher scores indicated positive coparenting.
Time Frame: 12 weeks postpartum
Population: Analysis population included only mothers who completed the scale at 12 weeks postpartum.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 100 | 96
units on a scale | 179.9 (27.4) | 174.9 (27.4)
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Breastfeeding Support
Description: Breastfeeding support is defined as the appraisal, emotional, informational and instrumental support the mother receives from her partner. This component of coparenting will be measured using the Postpartum Partner Support Scale (PPSS), which is a 24-item self-report instrument. The items are rated on a 4 point scale to produce a summative score ranging from 25-100. Two negative items are reversed scored and the higher scores indicate higher levels of postpartum-specific partner support.
Time Frame: 6 weeks
Population: Analysis population included only mothers who completed the scale at 6 weeks postpartum.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 98 | 91
units on a scale | 88.0 (10.9) | 85.6 (10.5)
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

8. Secondary Outcome: Breastfeeding Support
Description: as for outcome 7
Time Frame: 12 weeks
Population: Analysis population included only mothers who completed the scale at 12 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 100 | 96
units on a scale | 86.6 (11.7) | 83.6 (14.4)
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Paternal Breastfeeding Self-Efficacy
Description: Breastfeeding Self-Efficacy Scale- Short Form will be adapted and used to assess fathers' confidence with assisting their partner with breastfeeding.
  This instrument has 14 items, with responses ranging from 1-5. The total scores range from 14-70 with higher scores indicating higher breastfeeding self-efficacy.
Time Frame: 6 weeks postpartum
Population: Analysis population included fathers completed the scale and who had infants breastfeeding at 6 weeks postpartum (fathers of infants fed expressed breastmilk were not included).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 93 | 95
units on a scale | 55.9 (8.4) | 53.1 (11.2)
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

10. Secondary Outcome: Paternal Infant Feeding Attitude
Description: Paternal infant feeding attitude will be assessed using the Iowa Infant Feeding Attitude Scale. This scale consist of 17 items with a five point response range (1-5). The total scores range from 17-85. Negative items were reverse scored. Lower scores indicate a preference for formula feeding, while higher scores indicating a preference for breastfeeding.
Time Frame: 6 weeks postpartum
Population: Analysis population included only fathers who completed the scale at 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Number analyzed (Participants) | 93 | 95
units on a scale | 62.1 (8.1) | 61.2 (6.7)
Statistical Analysis 1: Comparison: Coparenting Breastfeeding Support Intervention vs Usual Care Group; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months data collection time period
Arm/Group | Coparenting Breastfeeding Support Intervention | Usual Care Group
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/214
Other Adverse Events (participants affected / at risk) | 0/214 | 0/214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No